CLINICAL TRIAL: NCT06632418
Title: A Randomized Controlled Trial Evaluating the Safety and Feasibility of the Recombinant Human Platelet-derived Growth Factor B (rhPDGF-BB)-Enhanced Collagen Plug for Complex Perianal Fistula Healing
Brief Title: Evaluating an rhPDGF-BB-enhanced Collagen Plug for Perianal Fistula Healing
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexander Hawkins (Other)
Collaborators: Lynch Regenerative Medicine, LLC (Unknown)
Responsible Party: Sponsor-Investigator, Alexander Hawkins, Director, Colorectal Research Center, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 240585
Record Dates: First submitted 2024-10-02; First posted 2024-10-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Anal Fistula; Complex Perianal Fistula
Keywords: Platelet-derived Growth Factor; Type 1 Collagen; Anal fistula plug
MeSH Terms: conditions — Rectal Fistula; Osteogenesis Imperfecta, Type IV | interventions — Becaplermin

STUDY DESIGN:
Intervention Model Description: Participants in the control arm of the study who have not healed by the time they reach the primary endpoint will have the option to crossover to the investigational arm and receive the investigational intervention. Their outcome measures will be tracked and documented, but their results will not be included in the initial analyses of the original randomized participant data. This will be considered extended open-label use of the investigational intervention and their outcome measures will be analyzed and reported separately.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Routine care (No Intervention): Participants receive routine care for their fistula.
- rhPDGF-BB-enhanced collagen plug (Experimental): Participants receive collagen plug saturated with rhPDGF-BB.
  Interventions: Drug: RhPDGF-BB

INTERVENTIONS:
Drug: RhPDGF-BB — 0.3 mg/mL rhPDGF-BB
  Arms: rhPDGF-BB-enhanced collagen plug

SUMMARY:
The average success rate for healing and remission of complex perianal fistulas, idiopathic or Crohn's-related, is approximately 50%. These abnormal connections between the rectum and the outside skin remain a major clinical challenge in need of new treatments aimed at tissue repair. Platelet-derived growth factor drives wound healing and tissue regeneration, and manufactured PDGF is currently used to heal diabetic foot ulcers and regenerate bone in periodontal and orthopedic patients. Manufactured recombinant human PDGF has the potential to improve the success rate for complete healing of complex perianal fistulas, reduce the recurrence rate due to reopening of the fistula tract, and avoid complications associated with routine surgical interventions.

DETAILED DESCRIPTION:
Perianal fistula is a common colorectal condition with an incidence of 9 cases per 100,000. Most perianal fistulas originate from an anal abscess that does not heal properly and are mainly treated with surgical interventions. The type of surgery and healing rates depend on the classification of the fistula as simple or complex and the proportion of the sphincter muscle that is involved. The second most common cause of perianal fistula is due to Crohn's disease (CD), a chronic inflammatory disease with an estimated annual incidence of 3 to 20 cases per 100,000. Approximately 20% of patients with CD will develop a perianal fistula within 10 years of diagnosis. CD-related perianal fistulas are a severe complication of chronic intestinal inflammation and rely on the combination of pharmacological therapies and surgical interventions, but still one-third of CD-related fistulas remain unhealed.

This Phase II clinical trial will evaluate the performance, preliminary safety and efficacy, and feasibility of the rhPDGF-BB-enhanced collagen plug versus routine care on healing complex perianal fistulas that are not eligible for a fistulotomy. This prospective, blinded, single-site study will randomize participants, 2:1 intervention versus control, into two arms comparing the rhPDGF-BB-enhanced collagen plug to routine care procedures and stratify participants by fistula etiology, Crohn's or idiopathic. Routine care includes draining seton removal and natural healing for Crohn's fistulas or COOK Biotech's Biodesign® Anal Fistula Plug implant for idiopathic fistulas. For both non-CD (idiopathic) and CD-related fistulas, a loose seton is an effective first-line treatment to facilitate drainage of the abscess, prevent the recurrence of an abscess, and increase the chance of healing successfully. After seton placement, the therapeutic interventions for idiopathic and CD-related fistulas differ, and the overall healing rates are widely variable in the literature. The outcomes for CD-related perianal fistulas with seton intervention report success rates between 14-81% and idiopathic perianal fistulas with anal fistula plug intervention are highly similar with success rates between 15.8-72.7%.

After recruiting and consenting, participants will be randomized and scheduled for the baseline procedure. Randomization blocks of size 3 (2:1 intervention to control) within each stratum (idiopathic versus CD-related) will be utilized, and the patient will be blinded. The investigator will not be blinded because the control and intervention procedures are different. Following the baseline procedure, participants will return for outcomes assessment by a blinded physician at one month, three months, and six months and complete a weekly participant survey from home. At each study visit, the blinded physician will perform a clinical examination of the external opening to assess for inflammation, drainage, and epithelialization, take clinical photographs, and discuss any adverse events (1-month and 3-month visits only). At the 3-month study visit, the blinded physician will determine if the fistula has completely healed, and this will be documented in the study database. At the 6-month final study visit, the blinded physician will assess for recurrence of the fistula by examination of the external opening, and this will be documented in the study database.

If the fistula is not healing at the 3-month study visit and the participant is in the control arm of the study, they will reach their endpoint as a control and have the option to crossover to the investigational arm and receive the investigational intervention. These participants will first have another draining seton placed in their fistula tract for approximately 3 weeks and be scheduled for the intervention procedure, implantation of the rhPDGF-BB-enhanced collagen plug. This group will restart at visit 2 for the procedure and return for all post-procedural study visits 3-5 at 1-, 3-, and 6-months. Their outcome measures will be tracked and documented, and they will complete the weekly participant surveys, but their results will not be included in the initial analyses of the original randomized participant data. This will be considered extended open-label use of the investigational intervention and will not delay reporting the outcomes from the comparison of healing between the original intervention and control groups at 3 months. Their outcome measures will be analyzed and reported separately.

The natural history and actual case-counts of these two patient populations, idiopathic and CD-related complex perianal fistulas, guided the design of the objectives, outcomes, and sample size that would allow this pilot study to be completed in approximately 15 months. A small, 2:1 randomized, parallel arm design was chosen for the purposes of evaluating preliminary performance, safety, efficacy, and feasibility. The primary objective of this study is to evaluate the technical performance of the rhPDGF-BB-enhanced collagen plug for the treatment of complex perianal fistulas regardless of etiology. This outcome measure is defined as procedural success of the rhPDGF-enhanced collagen plug without any intervention-related serious adverse events. Procedural complications include but are not limited to acute infection, dislodgement or extrusion of the plug, and non-healing of the fistula tract. The secondary objectives that are focused on the potential efficacy of this treatment will include a stratified subgroup analyses for idiopathic and CD-related fistulas due to the differences in natural history and potential differences in outcomes with routine care in these two groups. Further, the stratified, randomized design will promote balance of the etiologies across the trial arms. For this pilot, published data and the investigator's real-world experience with healing in these patients were used to design the objectives and outcomes that will guide a larger more definitive follow-up trial where assessing efficacy may or may not include both etiologies. Given the number of different perianal fistula types, anatomical presentations, and approaches to treatment, the inclusion criteria are specific to fistulas that are a single continuous tract, have had a draining seton placed, and are not amenable to fistulotomy regardless of etiology. The study design, control groups, and inclusion criteria support the endpoint analyses at 1-, 3-, and 6-months post intervention based on historical data for healing, remission, and recurrence of perianal fistulas.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a single tract perianal fistula not amenable to fistulotomy as determined by the supervising surgeon
* Fistula must currently have a draining seton in place
* Aged >21 years old
* Willing and able to provide informed consent and to comply with study protocol and follow-up
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Medical conditions that would, in the opinion of the investigator or treating provider, compromise the safety of the individual with study participation and/or the ability of the individual to follow study protocol
* Genito-urinary fistulization, including rectovaginal (i.e., fistulas that transverse the vaginal canal)
* Presence of an ileal anal pouch
* Any major surgery of the gastrointestinal tract (including one or more segments of the colon or terminal ileum) within 3 months prior to randomization; presence of stoma is not exclusionary
* Prior surgical procedure (i.e., Ligation of Intersphincteric Fistula Tract or Endorectal Advancement Flap) for the target fistula or a perianal procedure that resulted in a large soft tissue defect within 6 months prior to screening visit
* One or more of the following fistula types or anatomic presentations: horseshoe fistulas, fistulas that do not have an opening inside the anal canal or low rectum, blind ending sinus tracts (no external opening), branching fistulas (a previously performed conversion of a branching fistula tract to a single tract is not exclusionary), >1 internal opening, moderate or severe proctitis, severe rectal mucosal fibrosis surrounding the internal opening preventing the securing of the fistula plug disk, any anatomical limitation to successfully securing the fistula plug disk.
* Known allergic reactions to porcine collagen or yeast-derived products
* Currently enrolled in a drug or device trial or within 30 days of last investigational drug or device administration at baseline visit where investigational treatment (drug or device) was placed in or near the fistula tract or may potentially interact with study treatment
* Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
* Active infection at the application site
* The presence of malignant neoplasms at the application site
* Prior radiation therapy at the application site

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Without Treatment-Related Serious Adverse Events (SAEs) at 3 Months | Month 3
  Proportion of participants with procedural success as defined by implantation of the device without device-related SAEs.

SECONDARY OUTCOMES:
Number of Participants Who Achieved Fistula Healing at 3 Months | Month 3
  Fistula healing is a binary endpoint (healed or not healed) that will be determined by an evaluation from the blinded physician confirming whether there is visible drainage from the external opening.
Number of Participants With Fistula Recurrence at 6 Months | Month 6
  A participant that was diagnosed with a healed fistula that is diagnosed with recurrence of the fistula by clinical evaluation of the external opening at the 6-month follow-up visit.
Change from Baseline in Symptoms at Week 24 | From enrollment to week 24
  Weekly self-reported participant surveys assessing the prevalence of perianal fistula-related symptoms (including pain, incontinence, and missed days of school or work).
Change from Baseline in Pain on an 11-Point Scale at Week 24 | From enrollment to week 24
  Weekly self-reported participant surveys will be assessing average pain intensity through an 11-point scale. Possible scores range from 0 (No Pain) to 10 (Worst Pain).
Change from Baseline in Incontinence on a 5-Point Scale at week 24 | From enrollment to week 24
  Weekly self-reported participant surveys measuring incontinence with 5 questions (adapted from Wexner Incontinence Score) using a 5-point ordinal scale from 0 (Never) to 4 (Always (once or more per day)).
Number of Participants Recruited and Eligible | Monthly up to month 15
  Total number of participants that were recruited and eligible for the study.
Number of Participants Randomized Per Month | Monthly up to month 15
  Number of participants that were randomized each month of the study.
Proportion of Participants Retained at 3 and 6 Months | Month 3 and month 6
  Proportion of participants retained in the study at the 3 month and 6 month endpoints.
Summary of Device-Related Adverse Events (AEs) | Month 3
  A quantitative and descriptive summary of all device-related AEs. Relationship to study intervention will be assessed by the clinician who examines and evaluates the participant based on temporal relationship and his/her clinical judgment.

OTHER OUTCOMES:
Crossover Outcomes | Month 3
  The proportion of crossover participants that are completely healed at 3-months following the investigational procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Hawkins, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided